CLINICAL TRIAL: NCT05100498
Title: Web-based Oncofertility Support Tool for Reproductive-age Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chin-Tsung Shen, Mackay Medical College, Mackay Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSM/VGH-2019-12-009CC
Record Dates: First submitted 2021-10-07; First posted 2021-10-29 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Breast Neoplasm Female; Fertility Preservation
Keywords: breast cancer; fertility preservation; social support; Ottawa Decision Support Framework; website
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-based oncofertility support tool (Experimental): User-centered design practices were used to develop an oncofertility support website for women with breast cancer before treatment. The steps of the Ottawa Decision Support Framework were used throughout the development process. A multidisciplinary steering group was assembled, and the input was provided. Guidelines from the International Patient Decision Aid Standards were applied to test the quality of the oncofertility support website.
  Three steps included:
  1. Identify the supportive needs of a patient;
  2. Guide the development of support interventions;
  3. Evaluate the quality of web-based oncofertility support.
  Interventions: Device: Web-based oncofertility support tool

INTERVENTIONS:
Device: Web-based oncofertility support tool — The website structure was developed to satisfy the needs of reproductive-age women was investigated based on four domains of social support, as developed by Cohen and Syme (1985). The important needs of patients can be classified as emotional, informational, appraisal, and instrumental support.

SUMMARY:
The aim of this study was to develop electronic systems (e-systems) for oncofertility support, and to examine the comprehensibility, feasibility, usability, and effects on social support and preparation for decision-making.

DETAILED DESCRIPTION:
Background: When reproductive-aged women with breast cancer lack support in making decisions about fertility, this results in conflicts in decision-making with negative effects on their mental health.

Objective: The aim of this study was to develop electronic systems (e-systems) for oncofertility support, and to examine the comprehensibility, feasibility, usability, and effects on social support and preparation for decision-making.

Methods: The study steps were guided, tested, and utilized to (a) identify the requirements of a patient, (b) guide the development of support interventions, and (c) evaluate the quality of web-based oncofertility support. Both qualitative and quantitative data were collected to explore supportive requirements related to oncofertility care, and an initial website concerning oncofertility was developed based on the resulting requirements and system review regarding social support. Alpha testing and beta testing were used to ensure the quality of the web-based oncofertility support tool. The effectiveness was evaluated using the Preparation for Decision-Making Scale and Social Support Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Health provider who ever cared the patients with breast cancer.
* Patients with breast cancer aged between 20 and 45.

Exclusion Criteria:

* Patients of severe psychiatric disorders.
* Patients under 20 years old.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Degree of social support rated before and after using the web-based tool by patients | 4 months
  Social support was measured using a 16-item Likert-type questionnaire rating (from 0-3). Women of reproductive age were instructed to complete the social support questionnaire, assessing four dimensions of social support: emotional, informational, appraisal, and instrumental, before and after using the web-based tool.

SECONDARY OUTCOMES:
Preparation for Decision Making (PrepDM) evaluated by patients and healthcare providers | 4 months
  Both patients and healthcare providers were instructed to evaluate the Preparation for Decision Making Scale by the Joint Commission of Taiwan. All participants were instructed to respond to 10 questions based on a five-point Likert scale rating (from 1-5). A higher score indicates a greater agreement with the effect.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Miauh Huang, PhD, Principal Investigator — Department of Nursing
Locations (1):
- Department of Nursing, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang SM, Tseng LM, Yang MJ, Chang A, Lien PJ, Hsiung Y. Developing a web-based oncofertility tool for reproductive-age women with breast cancer based on social support framework. Support Care Cancer. 2022 Jul;30(7):6195-6204. doi: 10.1007/s00520-022-07046-x. Epub 2022 Apr 19. PMID 35438338
- See also: Web-based oncofertility support tool for reproductive-age women with breast cancer — https://sites.google.com/mmc.edu.tw/oncofertility/home